CLINICAL TRIAL: NCT05086796
Title: Substance Use Treatment and Recovery Team
Acronym: START
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: RAND (Other); University of New Mexico (Other); Baystate Health (Other); National Center for Advancing Translational Sciences (NCATS) (NIH); National Institute on Drug Abuse (NIDA) (NIH); Stanford University (Other); University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Itai Danovitch, Professor and Chair Department of Psychiatry & Behavioral Neurosciences, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000515; 5U01TR002756-02 (NIH); 1U01TR002756-01A1 (NIH)
Record Dates: First submitted 2021-10-12; First posted 2021-10-21 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Opioid-use Disorder; Opioid-Related Disorders
Keywords: Collaborative Care; Hospital; Addiction; Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Substance Use Treatment and Recovery Team (START) (Active Comparator): The intervention is administered to participants in this arm. Participants in this arm will work with the Substance Use Treatment and Recovery Team (START), a collaborative care team for inpatients with opioid use disorder.
  Interventions: Behavioral: Substance Use Treatment and Recovery Team (START)
- Usual Care (No Intervention): Usual care for people with opioid use disorder.

INTERVENTIONS:
Behavioral: Substance Use Treatment and Recovery Team (START) — START is a model of care based on Collaborative Care. START is team driven, population-focused, measurement based, and focused on promoting adoption of evidence-based interventions. The purpose of this model is to increase adoption of evidence-based interventions for opioid use disorder and to increase linkage to aftercare.
  The components of the START intervention are as follows:
  1. Triage
  2. Engage, Assess, and Plan
  3. Treat
  4. Communicate and Coordinate
  5. Follow up
  6. Monitor
  Arms: Substance Use Treatment and Recovery Team (START)

SUMMARY:
This study is a multi-site, randomized pragmatic trial being conducted at three diverse sites. The study, called the Substance Use Treatment and Recovery Team (START), will evaluate whether a collaborative care team increases the use of two interventions-medication for opioid use disorder (MOUD), and opioid use disorder (OUD) focused discharge planning-among hospitalized patients with OUD, and improves linkage to follow-up care relative to usual care. The START consists of an addiction medicine specialist and a care manager who will use evidence-based tools to decrease barriers to MOUD and engage patients with post-discharge OUD care. A total of 414 patients will be randomized from Cedars-Sinai Medical Center in Los Angeles, the University of New Mexico Hospital in Albuquerque, and Baystate Health in Springfield, Massachusetts to receive either START or usual care, stratifying by prior MOUD exposure and site.

DETAILED DESCRIPTION:
In the past decade, hospitalizations for OUD nearly doubled. Patients admitted to the hospital with an underlying OUD rarely receive evidence-based treatment for OUD while hospitalized. MOUD is not commonly initiated in the hospital, and patients are seldom linked to outpatient treatment after discharge. Hospitalized patients with OUD who do not initiate MOUD or receive linkage to post-discharge treatment are at high-risk of continued misuse, delays in care, future overdose and costly readmission. This study identifies the inpatient hospital stay as a key opportunity to initiate MOUD and link patients with follow-up care for OUD.

The Substance Use Treatment and Recovery Team (START) is an intervention that adapts the principles of collaborative care to the hospital setting. Prior studies have demonstrated the effectiveness of collaborative care in outpatient settings for patients with opioid and alcohol use disorders, and a series of reports have demonstrated the feasibility and potential efficacy of hospital based consultative teams for substance use disorders. START uses team based, multi-faceted interventions (ie: motivational interviewing, medication treatment, OUD-focused discharge planning), measurement-based care, and patient registries to increase delivery of evidence-based care. The goal of START is to facilitate initiation of MOUD during the inpatient stay and link patients to appropriate post-discharge care.

The START study is a multi-site, randomized trial that will evaluate the intervention improves MOUD initiation and linkage to follow-up care among hospitalized patients with OUD. A total of 414 patients will be randomized from three geographically diverse hospitals (Cedars-Sinai Medical Center in Los Angeles, the University of New Mexico Hospital in Albuquerque, and Baystate Health in Springfield, Massachusetts) to receive either START or usual care, stratifying by prior MOUD exposure and site. The study builds on a pilot randomized controlled trial conducted at Cedars-Sinai by testing the intervention at three geographically distinct locations, thus increasing generalizability.

If the aims of the research are achieved, the investigators will learn whether this model of care increases OUD treatment delivery in general medical hospitals, and decreases the downstream effects of untreated OUD. If effective, this translational model also can be used to increase uptake of evidence-based practices for other substance use and behavioral health disorders.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to an inpatient bed at Cedars-Sinai Medical Center (CSMC),University of New Mexico Hospital (UNM), or Baystate Health (BH)
* Age 18 and older
* Have a probable OUD diagnosis, defined by scores of > 3 on the opioid section of the Alcohol, Smoking, and Substance Involvement Screening test (ASSIST)
* Speaks English or Spanish as primary language
* Willing to participate in follow-up calls and interview by telephone and able to provide contact information for follow-up calls
* Able to provide informed consent

Exclusion Criteria:

* Currently receiving FDA-approved medication treatment for an opioid use disorder
* < 6 months life expectancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2023-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Itai Danovitch, MD, Principal Investigator — Cedars-Sinai Medical Center; Allison J Ober, PhD, Principal Investigator — RAND
Locations (3):
- United States (3):
  - Cedars Sinai Medical Center, Los Angeles, California
  - Baystate Medical Center, Springfield, Massachusetts
  - University of New Mexico Hospital, Albuquerque, New Mexico

IPD SHARING:
Plan to Share IPD: Yes
The data and associated documentation will be made available to users under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying the data after analyses are completed.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be available upon completion of analyses until five years after study completion.
Access Criteria: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying the data after analyses are completed.

REFERENCES:
- [Derived] Ober AJ, Murray-Krezan C, Page K, Friedmann PD, Anderson J, Osilla KC, Ryzewicz S, Huerta S, Mazer MW, Hoskinson RA, Garvey R, Peltz A, Watkins KE, Nuckols T, IsHak WW, Mariano LT, Danovitch I. Hospital Addiction Consultation Service and Opioid Use Disorder Treatment: The START Randomized Clinical Trial. JAMA Intern Med. 2025 Jun 1;185(6):624-633. doi: 10.1001/jamainternmed.2024.8586. PMID 40193131
- [Derived] Ober AJ, Murray-Krezan C, Page K, Friedmann PD, Chan Osilla K, Ryzewicz S, Huerta S, Mazer MW, Leamon I, Messineo G, Watkins KE, Nuckols T, Danovitch I. The Substance Use Treatment and Recovery Team (START) study: protocol for a multi-site randomized controlled trial evaluating an intervention to improve initiation of medication and linkage to post-discharge care for hospitalized patients with opioid use disorder. Addict Sci Clin Pract. 2022 Jul 28;17(1):39. doi: 10.1186/s13722-022-00320-7. PMID 35902888

RESULTS

PARTICIPANT FLOW:
Groups:
- Substance Use Treatment and Recovery Team (START): The intervention is administered to participants in this arm. Participants in this arm will work with the Substance Use Treatment and Recovery Team (START), a collaborative care team for inpatients with opioid use disorder.
  Substance Use Treatment and Recovery Team (START): START is a model of care based on Collaborative Care. START is team driven, population-focused, measurement based, and focused on promoting adoption of evidence-based interventions. The purpose of this model is to increase adoption of evidence-based interventions for opioid use disorder and to increase linkage to aftercare.
  The components of the START intervention are as follows:
  1. Triage
  2. Engage, Assess, and Plan
  3. Treat
  4. Communicate and Coordinate
  5. Follow up
  6. Monitor
Period: Overall Study
Arm/Group | Substance Use Treatment and Recovery Team (START) | Usual Care
Started | 164 | 161
Completed | 125 | 104
Not Completed | 39 | 57

BASELINE CHARACTERISTICS:
Population: Intention-to-treat population defined as all participants who met eligibility criteria, consented, and were randomized to one of the two treatment arms.
Groups:
- Total: Total of all reporting groups
Arm/Group | Substance Use Treatment and Recovery Team (START) | Usual Care | Total
Number analyzed (Participants) | 164 | 161 | 325
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 41.5 [34 to 50] | 40 [31 to 51] | 41 [32 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 48 | 112
  Male | 100 | 113 | 213
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 81 | 75 | 156
  Not Hispanic or Latino | 83 | 86 | 169
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 12 | 16 | 28
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 12 | 21
  White | 66 | 59 | 125
  More than one race | 10 | 13 | 23
  Unknown or Not Reported | 65 | 60 | 125
Region of Enrollment [Number; unit: participants]
  United States | 164 | 161 | 325

OUTCOME MEASURES:

1. Primary Outcome: In-hospital Initiation of MOUD Therapy
Description: Initiated MOUD prior to discharge, defined as use of any FDA-approved pharmacotherapy for OUD, including buprenorphine, naltrexone and methadone (Binary)
Time Frame: During the inpatient stay, an average of 7 days
Population: Intention-to-treat: All participants who met eligibility criteria and were randomized to one of the two arms.
Measure: Count of Participants; unit: Participants
Arm/Group | Substance Use Treatment and Recovery Team (START) | Usual Care
Number analyzed (Participants) | 164 | 161
Participants | 94 | 43
Statistical Analysis 1: Comparison: Substance Use Treatment and Recovery Team (START) vs Usual Care; Test type: Superiority; Risk Ratio (RR) = 2.10, 97.5% CI 2-sided [1.51 to 2.91] — The START arm is the numerator, Usual Care is the denominator. There are two primary outcome measures, so the type I error level was adjusted to alpha = 0.025; Poisson regression was used to compare the proportions of participants who initiated MOUD in the hospital by calculating the risk ratio (RR) and 97.5% confidence interval (CI) and with covariates treatment arm, site (3 sites), prior exposure to MOUD (yes vs. no), and length of hospital stay in days

2. Primary Outcome: Linkage to Follow-up OUD Care
Description: Attended at least one OUD-related care visit within 30 days of hospital discharge (Binary)
Time Frame: 30 days
Population: Intention-to-treat: All participants who met eligibility criteria and were randomized to one of the two arms and who had a follow-up visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Substance Use Treatment and Recovery Team (START) | Usual Care
Number analyzed (Participants) | 125 | 104
Participants | 90 | 50
Statistical Analysis 1: Comparison: Substance Use Treatment and Recovery Team (START) vs Usual Care; Test type: Superiority; Risk Ratio (RR) = 1.49, 97.5% CI 2-sided [1.15 to 1.93] — [estimate comment as in outcome 1, analysis 1]; Poisson regression was used to compare the proportions of participants who linked to follow-up OUD care by calculating the risk ratio (RR) and 97.5% confidence interval (CI) and with covariates treatment arm, site (3 sites), and prior exposure to MOUD (yes vs. no)

3. Secondary Outcome: OUD-specific Discharge Plan
Description: Received an after-hospital care plan that specifies a date and time for a post-discharge addiction care appointment (Binary)
Time Frame: During the inpatient stay, an average of 7 days
Population: Intention-to-treat: All participants who met eligibility criteria and were randomized to one of the two arms.
Measure: Count of Participants; unit: Participants
Arm/Group | Substance Use Treatment and Recovery Team (START) | Usual Care
Number analyzed (Participants) | 164 | 161
Participants | 81 | 44
Statistical Analysis 1: Comparison: Substance Use Treatment and Recovery Team (START) vs Usual Care; Test type: Superiority; Risk Ratio (RR) = 1.80, 95% CI 2-sided [1.35 to 2.41] — The START arm is the numerator, Usual Care is the denominator; Multivariable Poisson regression was used to compare the proportions of participants who initiated MOUD in the hospital between arms by calculating the risk ratio (RR) and 95% confidence interval (CI) with covariates: treatment arm, site (3 sites), and prior exposure to MOUD (yes vs. no)

4. Secondary Outcome: Any Post-discharge MOUD Utilization
Description: Initiated MOUD or continued MOUD treatment within 30 days following hospital discharge (Binary)
Time Frame: 30 days
Population: Intention-to-treat: All participants who met eligibility criteria and were randomized to one of the two arms and who had a follow-up visit and responded to this question.
Measure: Count of Participants; unit: Participants
Arm/Group | Substance Use Treatment and Recovery Team (START) | Usual Care
Number analyzed (Participants) | 124 | 104
Participants | 65 | 32
Statistical Analysis 1: Comparison: Substance Use Treatment and Recovery Team (START) vs Usual Care; Test type: Superiority; Risk Ratio (RR) = 1.71, 95% CI 2-sided [1.23 to 2.39] — The START arm is the numerator, Usual Care is the denominator; Multivariable Poisson regression was used to compare the proportions of participants who reported any post-discharge MOUD utilization between arms by calculating the risk ratio (RR) and 95% confidence interval (CI) with covariates: treatment arm, site (3 sites), and prior exposure to MOUD (yes vs. no)

5. Secondary Outcome: Post-discharge Outpatient Medical Care
Description: Completed at least one visit to an outpatient medical provider within 30 days of hospital discharge (Binary). Visit must be specifically related to opioid use and may include an emergency department visit.
Time Frame: 30 days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Substance Use Treatment and Recovery Team (START) | Usual Care
Number analyzed (Participants) | 122 | 104
Participants | 42 | 19
Statistical Analysis 1: Comparison: Substance Use Treatment and Recovery Team (START) vs Usual Care; Test type: Superiority; Risk Ratio (RR) = 1.89, 95% CI 2-sided [1.18 to 3.03] — The START arm is the numerator, Usual Care is the denominator; Multivariable Poisson regression was used to compare the proportions of participants who reported receiving any post-discharge outpatient medical care for their OUD between arms by calculating the risk ratio (RR) and 95% confidence interval (CI) with covariates: site (3 sites), and prior exposure to MOUD (yes vs. no)

6. Secondary Outcome: Past 30-day Number of Days With Any Opioid Use
Description: Days of use in the past 30 days after hospital discharge - Adapted National Survey of Drug Use and Health (NSDUH) (Continuous). "Use-days" range from 0 to 120 days with up to 30 days of use reportable for each of four opioid categories: pain medications excluding fentanyl, fentanyl, heroin/opium alone, heroin/opium mixed with another drug
Time Frame: 30 days
Population: Intention-to-treat: All participants who met eligibility criteria and were randomized to one of the two arms and who responded to the question.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Substance Use Treatment and Recovery Team (START) | Usual Care
Number analyzed (Participants) | 122 | 103
days | 0.0 [0.0 to 10.0] | 0.0 [0.0 to 14.0]
Statistical Analysis 1: Comparison: Substance Use Treatment and Recovery Team (START) vs Usual Care; Test type: Superiority; Incident rate ratio = 1.25, 95% CI 2-sided [0.64 to 2.43] — The START arm is the numerator, Usual Care is the denominator; Multivariable negative binomial regression with a log link function was used to compare opioid use-days between the two treatment arms by calculating the incident rate ratio (IRR) and 95% confidence interval (CI) with covariates: site (3 sites), prior exposure to MOUD (yes vs. no), and baseline opioid use days

ADVERSE EVENTS:
Time Frame: 90 days - from date of enrollment to end of follow-up period.
Arm/Group | Substance Use Treatment and Recovery Team (START) | Usual Care
All-Cause Mortality (participants affected / at risk) | 3/164 | 3/161
Serious Adverse Events (participants affected / at risk) | 4/164 | 3/161
Other Adverse Events (participants affected / at risk) | 1/164 | 0/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Substance Use Treatment and Recovery Team (START) (N=164) | Usual Care (N=161)
Necrotizing oft-tissue infection (NSTI) (Infections and infestations) | 1 (1) | 0 (0) — Led to death
(Investigations) | 2 (2) | 2 (2) — Led to death
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) — Led to death
Hospitalized (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Substance Use Treatment and Recovery Team (START) (N=164) | Usual Care (N=161)
Grievance (Social circumstances) | 1 (1) | 0 (0) — Subject grievance expressed during a call in an effort to conduct the follow-up interview.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-08-08): https://cdn.clinicaltrials.gov/large-docs/96/NCT05086796/Prot_001.pdf
  • Statistical Analysis Plan (2024-12-10): https://cdn.clinicaltrials.gov/large-docs/96/NCT05086796/SAP_002.pdf
  • Informed Consent Form (2022-06-22): https://cdn.clinicaltrials.gov/large-docs/96/NCT05086796/ICF_000.pdf